CLINICAL TRIAL: NCT00416689
Title: Determination of Utilities for Control of Chemotherapy-Induced Nausea or Vomiting
Brief Title: Nausea or Vomiting in Patients Who Are Receiving Chemotherapy for Breast Cancer or Lung Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-309801; U10CA031946 (NIH); CALGB-309801; CDR0000460041 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer; Lung Cancer; Nausea and Vomiting
Keywords: nausea and vomiting; pulmonary carcinoid tumor; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Nausea; Vomiting; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast or lung CA pt undergoing chemoTx
  Interventions: Procedure: assessment of therapy complications; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: assessment of therapy complications
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Understanding how nausea or vomiting caused by chemotherapy effects a patient's treatment decisions may help doctors plan better cancer treatment and may help patients live more comfortably.

PURPOSE: This clinical trial is studying nausea or vomiting in patients who are receiving chemotherapy for breast cancer or lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the contribution of nausea or vomiting to the overall importance for a current state of health in patients with breast or lung cancer undergoing chemotherapy.
* Determine the average importance for various emetic scenarios in these patients.
* Compare the importance of a specific level of chemotherapy-induced nausea or vomiting, defined by the Standard Gamble vs Morrow Assessment of Nausea and Emesis.
* Determine the feasibility of using a Standard Gamble technique in patients currently undergoing chemotherapy.

OUTLINE: This is a multicenter study. Patients are stratified according to history of chemotherapy-induced nausea or vomiting (yes vs no).

Patients undergo a structured interview over 1 hour by a trained interviewer at least 2½ weeks after initiation of the most recent course of chemotherapy and before the new course is administered. Patients complete a Functional Assessment of Cancer Therapy-General questionnaire and Morrow Assessment of Nausea and Emesis questionnaire during the interview. The trained interviewer also administers a Standard Gamble exercise during the interview, in which patients are instructed to imagine various amounts of nausea or vomiting as their current state of nausea and vomiting, and rank their importance to them. They are being asked to answer the question of whether they would choose to accept their current (imagined or real) state of nausea or vomiting or receive a medication that would result (with various probabilities) in either perfect health for 2 years or immediate death.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer or lung cancer
* Must be undergoing chemotherapy with each course lasting 3-6 weeks AND meets all of the following criteria:

  * Completed ≥ 1 course with ≥ 1 additional course planned
  * At least 2½ weeks since initiation of the most recent course of chemotherapy

PATIENT CHARACTERISTICS:

* Common Toxicity Criteria performance status 0-2
* Must have command of written and/or spoken English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast or lung cancer patients undergoing chemotherapy
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2000-04; Primary Completion 2003-03 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grunberg, MD, Study Chair — University of Vermont Medical Center